CLINICAL TRIAL: NCT07362550
Title: A Comparative Study of Monozygotic and Dizygotic Twins: Evaluating the Effects of a 12-Week Balanced Diet Intervention on Body Composition and Metabolic Parameters.
Brief Title: Effects of 12-Week Balanced Diet on Body Composition & Metabolic Parameters in Twins
Acronym: TWIN-BD12
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Qaisar Raza, Assistant Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniversityUVAS1
Record Dates: First submitted 2025-12-17; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adults
Keywords: Monozygotic; Dizygotic; Metabolic Parameters

STUDY DESIGN:
Intervention Model Description: Parallel, randomized, twin-pair controlled interventional study in which one twin from each monozygotic and dizygotic pair receives a 12-week WHO-aligned balanced diet while the co-twin continues habitual diet, with pre- and post-intervention assessments of body composition and metabolic parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual Diet (No Intervention): Control group will remain on habitual Diet.
- Balanced Diet (Experimental): 12-week culturally adapted WHO-aligned balanced diet emphasizing whole grains, lean proteins, healthy fats, fruits, and vegetables, individualized based on basal metabolic rate (BMR) and physical activity levels will be provided to interventional arm.
  Interventions: Other: Balanced Diet

INTERVENTIONS:
Other: Balanced Diet — 12-week culturally adapted WHO-aligned balanced diet emphasizing whole grains, lean proteins, healthy fats, fruits, and vegetables.
  Macronutrient composition: 45-65% carbohydrates, 20-35% fats, 10-20% protein. Individualized based on basal metabolic rate (BMR) and physical activity.
  Weekly counseling and monitoring through dietary recalls and photographic diaries. This intervention aims to assess the effects of a balanced diet on body composition and metabolic parameters in monozygotic and dizygotic twins.
  Arms: Balanced Diet

SUMMARY:
Twin study in Lahore will assess genetic vs. environmental effects on diet and metabolism. Over 12 weeks, monozygotic and dizygotic twins will follow a WHO-aligned balanced diet. Body composition, metabolic markers, and adherence will be measured. Monozygotic twins are expected to show greater similarity in response, clarifying personalized nutrition strategies in Pakistan.

DETAILED DESCRIPTION:
Background: Twin studies help separate genetic and environmental influences on diet and metabolic health. With rising obesity and metabolic disorders in Pakistan, there is no twin-based dietary intervention data. Filling this gap is essential for developing effective, evidence-based personalized nutrition strategies.

Hypothesis: The null hypothesis states that there will be no difference in dietary response or within-pair similarity between monozygotic and dizygotic twins. The alternative hypothesis suggests that monozygotic twins will show greater similarity in diet response and that the balanced diet will significantly improve metabolic outcomes.

Methodology: A 12-week randomized controlled trial will recruit Monozygotic and Dizygotic twins aged 18-60 years in Lahore, Pakistan. Participants of interventional group will follow a WHO-aligned balanced diet. Body composition, metabolic markers, and dietary adherence will be assessed at baseline and week 12.

Statistical Design: Analyses will be conducted in SPSS using paired t-tests for within-pair comparisons and independent t-tests for Monozygotic vs. Dizygotic differences. Effect sizes will be calculated, with significance set at p < 0.05.

Expected Outcomes: The study is expected to show that the balanced diet improves metabolic and body composition outcomes, with monozygotic twins displaying more similar responses than dizygotic twins. These findings will clarify genetic vs. environmental effects and support more targeted nutrition recommendations in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female twins aged 18-60 years.
* Confirmed zygosity (MZ or DZ) based on a validated twin zygosity questionnaire.
* Both twins willing to participate for the entire intervention period.
* Free from chronic diseases requiring specialized diets (e.g., type 1 diabetes, celiac disease).
* Not currently enrolled in another dietary or lifestyle intervention study.

Exclusion Criteria:

* Pregnant or lactating women.
* Use of lipid-lowering, glucose-lowering, or weight-loss medications in the past 3 months.
* Major gastrointestinal disorders or conditions affecting nutrient absorption.
* Unwillingness to follow individualized dietary counseling or complete study assessments.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2026-04-19 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Change in Body Fat Percentage (%) | Baseline and after 12-Week of Intervention.
  Change in total body fat percentage measured using the InBody analyzer to assess the effect of a 12-week balanced diet intervention.

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose (mg/dL) | Baseline and after 12 weeks
  Change in fasting plasma glucose concentration measured to assess the metabolic effect of the 12-week balanced diet intervention.
  Unit: mg/dL Tool: Venous blood sample, enzymatic laboratory method
Change in Lipid Profile (mg/dL) | Baseline and after 12 weeks
  Change in fasting serum lipid concentrations measured to assess metabolic response to the 12-week balanced diet intervention. Includes:
  Total Cholesterol (mg/dL) Low-Density Lipoprotein (LDL-C, mg/dL) High-Density Lipoprotein (HDL-C, mg/dL) Triglycerides (mg/dL) Unit: mg/dL Tool: Venous blood sample, standard enzymatic laboratory methods
To compare within-pair similarity of Dietary Response | Baseline and after 12-Weeks of intervention
  To compare the within-pair similarity of diet response between Monozygotic (MZ) and Dizygotic (DZ) twins, allowing estimation of genetic versus environmental contributions to dietary effects.

CONTACTS AND LOCATIONS:
Overall Officials: Qaisar Raza, Ph.D, Principal Investigator — UNIVERSITY OF VETERINARY AND ANIMAL SCIENCES, LHR.
Locations (1):
- University of Veterinary and Animal Sciences, Lhr., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No